CLINICAL TRIAL: NCT00572377
Title: Safety and Efficacy of Alprostadil (FemLife Gel) in the Treatment of Female Sexual Arousal Disorder
Brief Title: Alprostadil (FemLife Gel) in the Treatment of Female Sexual Arousal Disorder
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The investigator at Cedars stopped this study due to problems collecting payment from the sponsor.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Ernst Schwarz MD, Cedars Sinai Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB# 11268; FemLife
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Female Sexual Arousal Disorder
Keywords: Sexual; Arousal; Female
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FemLife Gel (Active Comparator)
  Interventions: Drug: FemLife Gel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FemLife Gel — the gel or placebo (240 mcg)applied to the vagina; 20 doses to be used over the 30 day period and to complete the Female Sexual Encounter Profile (FSEP).
  Arms: FemLife Gel
Drug: Placebo — the gel or placebo (240 mcg) applied to the vagina; 20 doses to be used over the 30 day period and to complete the Female Sexual Encounter Profile (FSEP).
  Arms: Placebo

SUMMARY:
Female sexual arousal disorder (FSAD) is a frequent finding in women in middle age and more prevalent in post-menopausal women. Topical alprostadil is currently under development for the treatment of FSAD. The purpose of this research is to determine if this formula of alprostadil is safe and effective in women with FSAD. We will be comparing alprostadil to placebo. Each participant will be treated for 1 month with active alprostadil and 1 month with placebo without knowing which they are using. This way, the investigators can compare the effects of alprostadil to the effects of an inactive topical gel.

Post-menopausal women with FSAD will be recruited. The women interested in participating in the study will first meet with investigators and answer questions to make sure they are eligible for the study and fit the diagnosis of FSAD.

Once enrolled, subjects will fill out questionnaires about their medical history, social history, and psychosocial history. They will also undergo medical examination. At this introductory research visit they will fill out baseline questionnaires, give medical history, undergo physical exam and have blood drawn. The informed consent will be reviewed and will be signed by the participant at this time.

The subject will then return for the 1st treatment visit at which time vital signs like blood pressure and heart rate will be taken, external genitalia will be examined and study drug will be dispensed after randomly being assigned to either alprostadil or placebo. After instruction, the subject will use first dose in the clinic and be monitored for 2 hours looking for changes in vital signs or local genitalia reaction. If no problems are noted, subject will be sent home with study drug and Female Sexual Encounter Profile Cards (FSEP). The patient will fill out these cards with each sexual encounter. After 1 week patient will be contacted by phone and asked about side effects or concerns. After 4 weeks the subject will return for another study visit at which time FSEP cards and left over study drug will be collected, questionnaires will be filled out, labs will be drawn and subject will undergo exam of external genitalia. The subject will then be sent home for a 2 week washout period.

The subject will return after this 2 week period with no study medication; she will then return and the above process will be repeated with either alprostadil or placebo (whichever she did not receive the first time).

ELIGIBILITY:
Inclusion Criteria:

1. FSAD based on American Foundation for Urological Disease Consensus Panel definition
2. Post-menopausal by WISE criteria or proof of bilateral oophorectomy.
3. FSAD for at least 6 months.
4. History of self reported normal sexual arousal and/or orgasm in the past.
5. Documentation of a normal PAP smear and pelvic exam within the past year.
6. Women may be on hormone replacement therapy because this is a non-hormonal therapy.

Exclusion Criteria:

1. Primary anorgasmia, vaginismus, sexual pain or sexual arousal disorder.
2. History of unresolved sexual trauma or abuse.
3. Endocrine disorders
4. Chronic UTI, vaginal infection, pelvic inflammatory disease, or dyspareunia within the preceding 12 months.
5. STI
6. Clinically significant renal, hepatic, neurologic, or cardiac disease in the preceding 6 months.
7. Male partner with impotence.
8. Depression or other mood disorder.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Female Sexual Encounter Profile (FSEP) | 30 days

SECONDARY OUTCOMES:
standardized questionnaire | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Schwarz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Mark Goodson Building, Los Angeles, California, United States

REFERENCES:
- [Background] 1. Basson R. Clinical practice. Sexual desire and arousal disorders in women. N Engl J Med. 2006;354:1497-506. 2. Addis IB et al. Reproductive Risk Factors for Incontinence Study at Kaiser Study Group. Sexual activity and function in middle-aged and older women. Obstet Gynecol. 2006;107:755-64. 3. Heiman JR et al. Topical alprostadil (PGE1) for the treatment of female sexual arousal disorder: in-clinic evaluation of safety and efficacy. J Psychosom Obstet Gynaecol. 2006;27:31-41 4. Kielbasa LA et al. Topical Alprostadil Treatment of Female Sexual Arousal Disorder Ann Pharmacother. 2006 Jun 6; [Epub ahead of print]. 5. Padma-Nathan H et al. Efficacy and Safety of Topical Alprostadil Cream for the Treatment of Female Sexual Arousal Disorder: A Double-Blind, Multicenter, Randomized, and Placebo-Controlled Clinical Trial. J of Sex and Marital Therapy. 29: 329-344, 2003.